CLINICAL TRIAL: NCT03849703
Title: Strengthening Relationships/Strengthening Families (SR/SF)
Brief Title: An Evaluation of Relationship and Coparenting Education Curricula for Adolescent Parents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Texas State University (Other)
Collaborators: Kansas State University (Other); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 90FM0067-01-01
Record Dates: First submitted 2018-03-06; First posted 2019-02-21 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Romantic Relationship Skills; Coparenting Skills
Keywords: Adolescent parents; coparenting; romantic relationships

STUDY DESIGN:
Intervention Model Description: An intent-to-treat randomized design coupled with a time-series design will be used to assess differential adjustment between the treatment and control groups, and to assess differential changes in adjustment between adolescent parents across four time-points. A block randomization design will be used to randomly assign eight participating schools into one of four treatment conditions based on curriculum assignment. Schools can receive a co-parenting (COPAR), healthy romantic relationship (HRR), and/or a control (CONT) curriculum each semester. Treatment conditions reflect schools which receive a full treatment model (i.e., COPAR-HRR, HRR-COPAR) or a partial treatment model (i.e., COPAR-CONT, and HRR-CONT).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Full Intervention #1 (Experimental): Participants will receive both of our target curricula but in alternate order. This treatment group will receive the coparenting curriculum before the romantic relationships curriculum.
  Interventions: Behavioral: Full Intervention #1
- Full Intervention #2 (Experimental): Participants will receive both of our target curricula but in alternate order. This treatment group will receive the romantic relationships curriculum before the coparenting curriculum.
  Interventions: Behavioral: Full Intervention #2
- Partial Intervention #1 (Other): Participants will receive the romantic relationships curriculum along with the control curriculum.
  Interventions: Behavioral: Partial Intervention #1
- Partial Intervention #2 (Other): Participants will receive the coparenting curriculum along with the control curriculum.
  Interventions: Behavioral: Partial Intervention #2

INTERVENTIONS:
Behavioral: Full Intervention #1 — Participants will receive 10 lessons on a weekly basis per semester for two semesters, for a total of 20 lessons. This Intervention group will receive the coparenting and then romantic relationship curricula. The lessons last between 45-60 minutes and are based on evidence based curricula.
  Arms: Full Intervention #1
Behavioral: Full Intervention #2 — Participants will receive 10 lessons on a weekly basis per semester for two semesters, for a total of 20 lessons. This Intervention group will receive the romantic relationship and then coparenting curricula. The lessons last between 45-60 minutes and are based on evidence based curricula.
  Arms: Full Intervention #2
Behavioral: Partial Intervention #1 — Participants will receive 10 lessons on a weekly basis per semester for two semesters, for a total of 20 lessons. This Partial Intervention group will receive the romantic relationship curriculum and a control curriculum. The lessons last between 45-60 minutes and are based on evidence based curricula.
  Arms: Partial Intervention #1
Behavioral: Partial Intervention #2 — Participants will receive 10 lessons on a weekly basis per semester for two semesters, for a total of 20 lessons. This Partial Intervention group will receive the coparenting curriculum and a control curriculum. The lessons last between 45-60 minutes and are based on evidence based curricula.
  Arms: Partial Intervention #2

SUMMARY:
An intent-to-treat randomized design coupled with a time-series design will be used to assess differential adjustment between the treatment and control groups, and to assess differential changes in adjustment between adolescent parents across four time-points. A block randomization design will be used to randomly assign eight participating schools into one of four treatment conditions based on curriculum assignment. Schools can receive a co-parenting (COPAR), healthy romantic relationship (HRR), and/or a control (CONT) curriculum each semester. Treatment conditions reflect schools which receive a full treatment model (i.e., COPAR-HRR, HRR-COPARE) or a partial treatment model (i.e., COPAR-CONT, and HRR-CONT). The investigators hypothesize that youth participating in the full-treatment group will show statistically significant immediate and sustained improvements in well-being, as well as larger improvements in their co-parenting and relationship knowledge and behaviors post treatment and more sustained improvements in co-parenting and relationship behaviors six months post-treatment than youth in the partial-treatment group. Couples in the program will show better co-parenting and relationship outcomes than couples where only one adolescent participated.

DETAILED DESCRIPTION:
Background The development of healthy romantic relationship skills and supportive co-parenting skills are important to family functioning and parental well-being. Family systems perspective and co-parental frameworks suggest these two relationships are related but distinct; however, curricula targeting family functioning do not target both relationship dynamics. A possible reason for this oversight may be that co-parenting curricula have been created for adult couples (e.g., Bringing Baby Home, Family Expectations, Family Foundations, Two Families Now; National Registry of Evidence-Based Programs and Practices [NREPP]). Similarly, healthy relationship programs have been targeted towards adolescents and emerging adults, or premarital couple where co-parenting was not given substantial attention.

Only two co-parenting curricula exist that target adolescent parents, the Young Parenthood Program (YPP) and the Family Foundations program (FFP). YPP states that it targets co-parenting skills, but the material actually targets healthy romantic relationship skills and the prevention of intimate partner violence (IPV), acknowledging youth developmental need to learn healthy relationship skills, but ignoring the saliency of co-parenting in this unique context. FFP does target the co-parenting relationship by focusing on identifying childrearing goals and duties and supporting the co-parental relationship; however, this program does not target healthy relationship dynamics or the prevention of IPV.

Unfortunately, adolescent parents, who are experiencing an off-time transition into early parenthood, face the challenge of learning to positively engage in romantic and co-parental relationships at the same time. To better serve this population, the Strengthening Relationships/ Strengthening Families (SR/SF) program is targeting healthy relationship and supportive co-parenting skills. Because a program targeting both skills has not been implemented in any population, our evaluation will move the field forward by showcasing the efficacy of targeting two family relationship dynamics concurrently. Further, by comparing a full-treatment (co-parenting and healthy relationships) to partial-treatment groups (co-parenting only or healthy relationship only), the investigators will be able to identify which relationship is more salient and impactful in increasing adolescent (e.g., depression, self-esteem, role overload) and parental (e.g., parental stress, parental self-efficacy) adjustment during this off-time transition into parenthood. Finally, cost-effectiveness analysis will also provide information of the program impacts if services are provided to one or both members of the co-parental system. Taken together, the program model and supporting evaluation will help build our knowledge of the most salient needs of adolescent parents, and program service delivery best practices.

Evaluation Questions and Hypotheses

Due to the lacuna in the literature focused on adolescent parents and their coparenting adjustment, the following research questions have been formulated:

1. Do pregnant and parenting adolescents who participate in the full-treatment group (Co-parenting AND Healthy Relationships) show larger improvements in their co-parenting and relationship knowledge and behaviors compared to those adolescents who participate in the partial-treatment group (Co-parenting OR Healthy Relationships)? H1: Youth participating in the full-treatment group will show larger improvements in their co-parenting and relationship knowledge and behaviors post treatment compared to youth in the partial-treatment group.
2. Do pregnant and parenting adolescents who participate in the full-treatment group show sustained improvements in co-parenting and relationship behaviors six-months post-treatment? H1: Youth participating in the full-treatment group will show more sustained improvements in co-parenting and relationship behaviors six months post-treatment than youth in the partial-treatment group.
3. Do couples who participate show significantly better co-parenting and relationship outcomes than couples where only one adolescent participated? (cost-effectiveness analysis) H1: Couples in the program will show better co-parenting and relationship outcomes than couples where only one adolescent participated.
4. Do pregnant and parenting adolescents who participate in the full-treatment group show immediate (post-treatment) and sustained (3- & 6-month follow-up) improvements in well-being (i.e., reduced depressive symptoms, role overload, increased parental self-efficacy)? H1: Youth participating in the full-treatment group will show statistically significant immediate and sustained improvements in well-being.

Impact Evaluation An intent-to-treat randomized design coupled with a time-series design will be used to assess differential adjustment between the treatment and control groups, and to assess differential changes in adjustment between groups across four time-points. SR/SF participants will be recruited to participate in this evaluation (See Sample Section below). In addition, non-SR/SF participant adolescent fathers will be recruited to participate in the evaluation to serve as a non-random control group. The time-series design will be administered pre-treatment (early Fall semester: August), mid-treatment (end of Fall semester: December; participants only), post-treatment (end of Spring semester: May), and three-months post-treatment (August). Each school year, data will be collected from a new cohort of participating pregnant/parenting adolescents (nparticipant/cohort = 160-200) and non-intervention fathers (nnon-participant/cohort = 40-50) for a total of four cohorts (nparticipant = 640-800; nnon-participant = 160-200).

Sample All students participating in our program beginning Fall 2016 will be invited to participate in this evaluation with the primary unit of analysis being the adolescent parent. The investigators will recruit 160-200 students/year for a total of 640-800 participants across four years. Our program participants are projected to be primarily female (75%), Hispanic (91%), pregnant and parenting (32% pregnant, 78% parenting) adolescents between the ages of 14-20, with an additional 40 adolescent fathers/year recruited (by the evaluation team) to serve as the non-equivalent control group for Research Question #3. Regardless of group membership, 440-550 adolescents will receive the co-parenting curriculum, and 440-550 adolescents will receive the healthy romantic relationship curriculum. Given our previous success in sample retention, less than 20% attrition is expected. However, our intent-to-treat design and missing data handling techniques will allow us to use the full sample in our analyses.

ELIGIBILITY:
Inclusion Criteria:

* pregnant or parenting (biological and nonbiological parents)
* adolescents

Exclusion Criteria:

-

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 640 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-09-29 (Estimated)

PRIMARY OUTCOMES:
Attitudes & Knowledge | 1 year
  The HMRE nFORM pre- and post-test surveys will be used to assess changes in attitudes towards marriage (Section A1), healthy relationships (Section A3), romantic relationship conflict resolution (Section A4), and intimate partner violence (Section A5).
Romantic Relationship Adjustment - Conflict Resolution | 1 year
  Abusive behaviors between dating adolescents will be assessed using the Conflict in Adolescent Dating Relationships Inventory (CADRI; Wolfe et al., 2001). Physical, sexual, emotional, verbal, and threatening behaviors are assessed in this 31-item measure. The CADRI has demonstrated acceptable test-retest reliability, good internal consistency, and agreement between dating partners (Wolfe, et al., 2001).
Coparenting Adjustment - Communication | 1 year
  Two subscales from the Co-parental Communication Scale (Ahrons, 1981) will be used to assess frequency of communication (7-item) and degree of conflict (7-item) that is present when discussing parenting issues between co-parents. This scale has been modified and validated with Mexican adolescent mothers (Madden-Derdich, 2002; Herzog, Umaña-Taylor, Madden-Derdich, & Leonard, 2007) with good reliability in both subscales (α > .78).

SECONDARY OUTCOMES:
Parenting - Involvement | 1 year
  Using the Parental Involvement Scale, parents will be asked to rate how frequently (4-point) they, the other biological parent, and their mothers engage in three types of activities with their infants: literacy, caregiving, and warmth (Cabrera, Shannon, & La Taillade, 2009). Having data on the target adolescent, the other parent, and mother, will allow us to assess parental and coparental involvement among families of adolescent parents. Previous work with Hispanic parents has shown good reliability (α =.87).
Psychosocial functioning - Self-esteem | 1 year
  Global self-esteem will be assessed using the 10-item Rosenberg Self-Esteem Scale (Rosenberg, 1979), which has been validated within Hispanic adolescent samples with good reliability (α >.71; Umaña-Taylor & Updegraff, 2007; Umaña-Taylor et al., 2004).

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03849703/Prot_SAP_000.pdf